CLINICAL TRIAL: NCT04194736
Title: Evaluation of the Occurrence of Early Thrombosis on Central Venous Catheter by Ultrasound in Pediatric Intensive Care Unit
Acronym: Thromb-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191078; 2019-A02893-54 (Other: IDRCB number)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Central Venous Catheters
Keywords: Percutaneous central venous catheter; Thrombosis; Children; Ultrasound scan
MeSH Terms: conditions — Thrombosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children (Experimental): Minor patients hospitalized in pediatric intensive care unit having a percutaneous central venous catheter.
  Interventions: Other: Ultrasound scan

INTERVENTIONS:
Other: Ultrasound scan — First ultrasound scan from 1 day to 6 days after the placement of the percutaneous central venous catheter.
  Second ultrasound scan from 7 days to 13 days after the placement of the percutaneous central venous catheter if no thrombosis was detected at the first ultrasound scan.

SUMMARY:
The objective of this study is to prospectively describe the incidence of early venous thrombosis secondary to the placement of a percutaneous central venous catheter, in a pediatric intensive care unit, by systematic ultrasound screening.

DETAILED DESCRIPTION:
In pediatric resuscitation, the use of a percutaneous central venous catheter is essential. It allows to administer strong osmolarity intravenous drugs or prolonged duration treatment and to carry out blood samples.

In the course of the placement of a central venous catheter, there is a risk of occurrence of early thrombosis between 20 and 45%, appearing mainly in the 4 first days. The occurrence is explained by the Virchow triad: endothelial lesion (linked to the central venous catheter), venous stasis, hypercoagulability. Ultrasonography is an imaging test that can be performed at the bedside, allowing the non-invasive collection of diagnostic elements of thrombosis (visible thrombus, non-compressibility of the vein, abolition of venous flow). Performing ultrasound for thrombosis screening is essential because of a very low clinical expression of thrombosis, while the consequences are potentially severe, including infection, embolism, venous insufficiency and loss of venous access for children who will need several central venous catheters during their lifetime.

Despite the knowledge of certain risk factors (i.e. assisted ventilation, history of cancer, transfusions,...), there is actually no consensus for the systematic screening of venous thromboses on central venous catheters. Systematic thromboprophylaxis is not recommended for central venous catheters (grade 1B). Concerning the curative treatment of central venous catheter thrombosis, unfractionated heparin or low molecular weight heparin (grade 1B) is recommended. If the central venous catheter is no longer needed for the care, it can be removed after 3 to 5 days of anticoagulants (grade 2C). It can also be kept under cover of anticoagulant treatment if its use is essential (grade 2C).

The objective of this study is to prospectively describe the incidence of early venous thrombosis secondary to the placement of a percutaneous central venous catheter, in a pediatric intensive care unit, by the systematic ultrasound screening.

ELIGIBILITY:
Inclusion Criteria:

- All children hospitalized in pediatric intensive care unit requiring the placement of a central venous catheter.

Exclusion Criteria:

* Impossibility of delivering an information in order to obtain a non-opposition.
* Absence of acoustic window (dressings).
* Removal of the catheter before performing the ultrasound.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence of the occurrence of thrombosis | Until 13 days after the placement of the percutaneous central venous catheter
  Occurrence rate of thrombosis.

SECONDARY OUTCOMES:
Risk factors for thrombosis | Until 13 days after the placement of the percutaneous central venous catheter
  Significant association between diagnosed thrombosis and risk factors, using univariate and multivariate analysis.
Time of onset of thrombosis | Until 13 days after the placement of the percutaneous central venous catheter
  Number of days between the catheter placement and the occurrence of thrombosis.
Therapeutic consequences of a thrombosis diagnosis | Until 13 days after the placement of the percutaneous central venous catheter
  Anticoagulant treatment or/and catheter removal.

CONTACTS AND LOCATIONS:
Overall Officials: Agathe Béranger, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No